CLINICAL TRIAL: NCT00425048
Title: Does Gloved Medical Personnel Scratch Less Often?
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Other Study IDs: A_B_19_01_2007
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Hygiene; Equipment Contamination; Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: wearing gloves

SUMMARY:
Unconscious touching of a person's own head or neck (for example by scratching) is a frequently observed and completely normal physiological movement pattern in humans, which when done by medical personnel attending a patient poses a high risk of unconscious self-contamination, even of an already disinfected hand, and of subsequent contamination of the patient. However, as compared to an ungloved hand, a gloved hand is felt to be "foreign," which could reduce the frequency of self-contact and thus the contamination rate.

Wearing protective gloves is highly recommended in medical practice. The purpose of this study is to explore how wearing, or not wearing, protective gloves affects

* the frequency of unconscious self-contact
* contamination of the gloved/ungloved hand

ELIGIBILITY:
Inclusion Criteria:

* Medical students working in a simulated OR environment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Benzer, MD, Principal Investigator — MUI Innsbruck
Locations (1):
- University Hospital, Innsbruck, Austria